CLINICAL TRIAL: NCT03688152
Title: A Phase 1b, Multicenter, Open-Label Study of the Safety and Tolerability of INCB053914 in Combination With INCB050465 in Participants With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: A Safety and Tolerability Study of INCB053914 in Combination With INCB050465 in Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 53914-102
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Relapsed Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma
Keywords: Diffuse large B-cell lymphoma; DLBCL; Non-Hodgkin lymphoma; phosphatidylinositol 3-kinase delta inhibitor; PI3Kδ; PIM kinases
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — parsaclisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INCB053914 + INCB050465 (Experimental): INCB053914 in combination with INCB050465.
  Interventions: Drug: INCB053914; Drug: INCB050465

INTERVENTIONS:
Drug: INCB053914 — Dose Escalation: INCB053914 at the protocol-defined starting dose in combination with INCB050465, with dose modifications based on tolerability criteria.
  Dose Expansion: Recommended dose from the dose-escalation study.
Drug: INCB050465 — Dose Escalation: INCB050465 at the protocol-defined starting dose in combination with INCB053914, with dose modifications based on tolerability criteria.
  Dose Expansion: Recommended dose from the dose-escalation study.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of INCB053914 in combination with INCB050465 in relapsed or refractory diffuse large B-cell lymphoma (DLBCL).

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory DLBCL, which has been histologically documented, defined as having received at least 2 but no more than 5 prior systemic treatment regimens (eg, an anti-CD20 antibody, an anti-CD20 antibody with or without chemotherapy, or chemotherapy alone) and ineligible for further treatment with standard of care.
* Willing to undergo pretreatment and on-treatment incisional or excisional biopsy of nontarget adenopathy or extranodal lesions. Provision of the most recent, available archived tumor biopsy may satisfy the pretreatment biopsy.
* Measurable disease as defined by the Lugano classification criteria:

  * ≥ 1 measurable nodal lesion (≥ 1.5 cm in longest dimension) or ≥ 1 measurable extranodal lesion (> 1 cm in longest dimension) on CT scan or MRI
  * ≥ 1 PET-avid lesion.
* Eastern Cooperative Oncology Group performance status 0 to 2.
* Willingness to avoid pregnancy or fathering children based on protocol-defined the criteria.

Exclusion Criteria:

* Laboratory values outside the protocol-defined range at screening unless approved by the medical monitor.
* Primary mediastinal (thymic) large B-cell lymphoma or Richter's Syndrome.
* Known brain or central nervous system metastases or history of uncontrolled seizures.
* Radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 2 weeks of the first dose of study treatment.
* Allogeneic stem cell transplant within the last 6 months, or active graft-versus-host disease following allogeneic transplant, or autologous stem cell transplant within the last 3 months before the date of the first dose of study treatment.
* Use of immunosuppressive therapy following allogenic transplant within 28 days of the first dose of study treatment.
* Prior treatment with a PIM inhibitor, selective PI3Kδ inhibitor (eg, idelalisib), or a pan-PI3K inhibitor.
* Receipt of anticancer medications, therapies, or investigational drugs within protocol-defined intervals before the date of the first dose of study treatment.
* Current or previous other malignancy within 3 years of study entry, except cured (or treated with curative intent and no evidence of disease) basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy without sponsor approval.
* History of liver function abnormality requiring investigation and/or treatment (eg, due to excessive alcohol or drug-induced liver injury).
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral, or psychiatric disease.
* Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment, and exposure to a live vaccine within 30 days of study treatment administration.
* Known HIV infection.
* Evidence of HBV or HCV infection.
* History of stroke or intracranial hemorrhage within 6 months of the date of study treatment administration.
* History of clinically significant or uncontrolled cardiac disease.
* Presence of an abnormal ECG that is clinically meaningful. Screening QTc interval > 480 milliseconds is excluded (corrected by Fridericia).
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study treatment and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events (TEAEs) | Up to approximately 6 months
  TEAE is defined as an adverse event reported for the first time or worsening of a pre-existing event after the first dose of study treatment.

SECONDARY OUTCOMES:
Cmax of INCB053914 in combination with INCB050465 | Day 15
  Maximum observed plasma concentration.
Tmax of INCB053914 in combination with INCB050465 | Day 15
  Time to maximum plasma concentration.
Cmin of INCB053914 in combination with INCB050465 | Day 15
  Minimum observed plasma concentration during the dosing interval.
AUC0-t of INCB053914 in combination with INCB050465 | Day 15
  Area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration.
Cl/F of INCB053914 in combination with INCB050465 | Day 15
  Oral dose clearance.
Overall response rate | Up to approximately 6 months
  Defined as the percentage of participants with a complete remission (CR)/complete metabolic response (CMR) or partial remission (PR)/partial metabolic response (PMR) as defined by investigator assessment per revised Lugano classification criteria for lymphomas.
Duration of response | Up to approximately 6 months
  Defined as the time from first documented evidence of CR/CMR or PR/PMR until disease progression or death from any cause among participants who achieve an objective response, as determined by radiographic disease assessment.
Progression-free survival | Up to approximately 6 months
  Defined as the time from the date of the first dose of any study drug until the earliest date of disease progression, as determined by radiographic disease assessment, or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Fred Zheng, MD, Study Director — Incyte Corporation
Locations (3):
- United States (3):
  - University of Arizona Cancer Center, Tucson, Arizona
  - UCLA Healthcare Hematology-Oncology, Santa Monica, California
  - Clinical Research Alliance, Lake Success, New York

IPD SHARING:
Plan to Share IPD: No